CLINICAL TRIAL: NCT04393779
Title: Beating Heart Mitral Valve REPair With the HARPOON™ System: ReaL World Outcomes From a multICenter observATional European Registry
Brief Title: Observational Registry on the HARPOON Device
Acronym: REPLICATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Edwards Lifesciences (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-12
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Results first posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Severe Degenerative Mitral Regurgitation Due to Mid-segment Posterior Leaflet Prolapse
Keywords: Mitral valve; Mid-segment posterior leaflet prolapse of the mitral valve; Heart valve; Chordae tendinae; Valve disease; Mitral Regurgitation; Harpoon; Mitral valve repair; Posterior leaflet prolapse; Beating heart intervention; Heart disease; Cardiovascular disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- HARPOON™ MVRS (Other): Subjects who were treated with the HARPOON MVRS.
  Interventions: Device: HARPOON Beating Heart Mitral Valve Repair System (MVRS)

INTERVENTIONS:
Device: HARPOON Beating Heart Mitral Valve Repair System (MVRS) — Repair of the chordae tendinae in the mitral valve.

SUMMARY:
To collect data on the HARPOON™ Mitral Valve Repair System for use in patients with severe degenerative mitral regurgitation due to posterior leaflet prolapse.

DETAILED DESCRIPTION:
This is a single arm, prospective, multicenter, post-market, observational registry that will evaluate subjects for up to 5 years post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are clinically suitable for treatment with the HARPOON™ System, as per the Instructions for Use (IFU), will be evaluated for inclusion in the registry.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walther, Prof Dr med, Principal Investigator — Goethe University
Locations (7):
- Germany (5):
  - Universitätsklinik Ulm, Ulm, Baden-Wurttemberg
  - Rhön Klinikum Kardiochirurgie, Bad Neustadt an der Saale, Bavaria
  - Klinikum Passau, Passau, Bavaria
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - Helios Universitätsklinikum Wuppertal, Wuppertal, North Rhine-Westphalia
- Hospital Son Espases, Palma, Balearic Islands, Spain
- Insel Gruppe AG, Universitätsklinik für Kardiologie, Schweizer Herz- und Gefässzentrum Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HARPOON™ MVRS
Started | 26
Completed | 21
Not Completed | 5
Not completed — Death | 1
Not completed — Device reintervention or explant | 4

BASELINE CHARACTERISTICS:
Arm/Group | HARPOON™ MVRS
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Re-operation Due to Recurrent Severe Mitral Regurgitation Through 1-year Post-implant
Description: Subject's freedom from re-operation due to recurrent severe mitral regurgitation through 1-year post-implant
Time Frame: 1 year post-implant
Population: This outcome is reported as a Kaplan Meier estimate for subjects who were attempted to be treated in the trial where data is available. The number of participants analyzed at the 1-year timepoint is equivalent to the number of patients at risk at that timepoint.
Measure: Number; unit: Percent of participants
Arm/Group | HARPOON™ MVRS
Number analyzed (Participants) | 15
Percent of participants | 81.0

ADVERSE EVENTS:
Time Frame: Adverse events occurring from baseline through 25 months post implant of the enrolled cohort.
Arm/Group | HARPOON™ MVRS
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 6/26
Other Adverse Events (participants affected / at risk) | 2/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HARPOON™ MVRS (N=26)
ACCESS SITE AND VASCULAR COMPLICATIONS - DAMAGE TO THE NATIVE MITRAL VALVE APPARATUS - CHORD (Vascular disorders) | 1 (1)
BLOOD SEPSIS (Blood and lymphatic system disorders) | 1 (1)
REGURGITATION - RECURRENT MITRAL SEVERE (Cardiac disorders) | 4 (4)
DEVICE SPECIFIC COMPLICATION - OTHER CHORD/KNOT PROBLEMS (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HARPOON™ MVRS (N=26)
REGURGITATION - RECURRENT MITRAL MODERATE (Cardiac disorders) | 1 (2)
DEVICE SPECIFIC COMPLICATION - OTHER CHORD/KNOT PROBLEMS (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can't publish/present on overall study results not yet published but may publish his own data subject to EW review prior to submission/presentation to ensure proprietary information shall not be divulged. Publication/presentation of the PI's site-specific results of devices which haven't been market released and which still may be undergoing development, shall not include claims of device safety/effectiveness and will require the review/approval of EW.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT04393779/Prot_SAP_000.pdf